CLINICAL TRIAL: NCT06999837
Title: [68Ga]Ga-PSMA PET/CT in Hepatocellular Carcinoma: Impact of Multiparametric Dynamic Whole-body Imaging and Kinetic Modeling.
Acronym: HIMIKO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC24_0482; 2024-515178-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-15; First posted 2025-05-31 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: HCC - Hepatocellular Carcinoma
Keywords: 68Ga-PSMA PET/CT; Hepatocellular carcinoma; multiparametric dynamic whole-body imaging
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [68Ga]Ga-PSMA (Experimental): Dynamic whole-body [68Ga]Ga-PSMA acquisition to HCC patients
  Interventions: Radiation: [68Ga]Ga-PSMA-11

INTERVENTIONS:
Radiation: [68Ga]Ga-PSMA-11 — Dynamic whole-body [68Ga]Ga-PSMA acquisition to HCC patients

SUMMARY:
The purpose of this study is to evaluate the use of multiparametric dynamic whole-body [68Ga]Ga-PSMA PET/CT imaging in newly diagnosed HCC patients or in HCC patients with recent suspicion of refractory, residual, or recurrent disease.

ELIGIBILITY:
Inclusion Criteria:

1. Provided written informed consent
2. Patient aged ≥ 18 years
3. For cohort A: patient with HCC histologically proven or who meet radiological criteria and are scheduled for biopsy For cohort B: patient with known HCC requiring a new diagnostic imaging workup for suspected refractory, residual or recurrent disease
4. Presence of at least one morphological evaluable lesion according to mRECIST 1.1 using contrast CT/MRI
5. Patient must have an ECOG (Eastern Cooperative Oncology Group) performance status of 0 to 2
6. Patient who are Child-Pugh A
7. Patient must have a life expectancy ≥ 6 months as determined by the study investigator
8. Patient affiliated to or beneficiary of the National Health Service
9. Consent to practice double-barrier contraception after [68Ga]Ga-PSMA injection (6 months of contraception for women study participant and their partners, and 3 months for men study participant and their partners)

Exclusion Criteria:

1. Known hypersensitivity to PSMA-11, to any excipient or derivative or to radiographic contrast agents
2. Patient requiring emergent surgery for a ruptured / bleeding HCC
3. Radioembolization within 3 months prior to inclusion
4. Cardiac disease with New York Heart Association classification of III or IV
5. Any major surgery within 4 weeks before enrollment
6. Other known malignancies (except for fully-resected non-melanoma skin cancer or cervical cancer in situ) unless definitively treated and proven no evidence of recurrence for 2 years
7. Any uncontrolled significant medical, psychiatric or surgical condition (active infection (subjects with known human immunodeficiency virus (HIV) positive)), unstable angina pectoris, cardiac arrhythmia, poorly controlled hypertension, poorly controlled diabetes mellitus (glycated haemoglobin (HbA1c) ≥9%), uncontrolled congestive heart disease, etc.) or laboratory findings that, in the opinion of the investigator, might jeopardise the subject's safety or that would limit compliance with the objectives and assessments of the study
8. Woman who are pregnant or breastfeeding. A serum pregnancy test will be performed at the start of the study for all female subjects of childbearing potential
9. Patient under guardianship or trusteeship
10. Patient under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-09-23 (Estimated); Study Completion 2027-09-23 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance | 6 months
  Sensitivity of qualitative assessment of dynamic whole-body [68Ga]Ga- PSMA PET/CT using standard imaging methods, pathological data if available data or imaging follow-up of at least 6 months as gold standard in two populations of HCC patients: at the time of initial diagnosis or upon detection of suspected refractory, residual, or recurrent relapse.

SECONDARY OUTCOMES:
Kinetic parameters | Baseline
  Patlak's parametric reconstruction, which estimates the 68 Gallium blood input function from the image, will be employed to extract the Ki absorption coefficient.
Diagnostic performance of multiparametric image evaluation approach at the lesion level | 6 months
  Sensitivity value of D-WB [68Ga]Ga-PSMA PET/CT and gold standard will be calculated and compared at the lesion level.
Diagnostic performance of multiparametric image evaluation approach at the patient level | 6 months
  Sensitivity value of static [68Ga]Ga-PSMA PET/CT and Choline-PET will be calculated and compared.
Diagnostic performance of multiparametric image evaluation approach at the patient level | 6 months
  Sensitivity value of dynamic [68Ga]Ga-PSMA PET/CT and Choline-PET will be calculated and compared.
Acceptability in terms of comfort | Baseline
  Acceptability will be measured by a comfort scale from 1 (very uncomfortable) to 5 (very comfortable).
Dynamic compared to static imaging | Baseline
  Target-to-background ratios (TBR) values were compared with Tumor normalized uptake values (SUV images) to evaluate lesions detection.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - HU Paris Nord APHP, Clichy
  - CHU de Nantes, Nantes

IPD SHARING:
Plan to Share IPD: Undecided